CLINICAL TRIAL: NCT00767273
Title: Pilot Study to Investigate the Role of Metabolic Imaging in Predicting Tumor Response and Outcome After Therapy for Pancreatic Cancer
Brief Title: Investigate Role of Metabolic Imaging in Predicting Tumor Response/Outcome After Pancreatic CA Tx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Albert Koong, Associate Professor of Radiation Oncology, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PANC0004; 95733; SU-11052007-795 (Other: Stanford University)
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: PET Scan
Drug: FLT
Drug: FDG

SUMMARY:
To test the ability of new imaging techniques to monitor and predict response of pancreatic cancer to radiation and/or chemotherapy.

ELIGIBILITY:
Inclusion Criteria:- Adult patients (>18) with histologically confirmed adenocarcinomas of the pancreas with a - treatment plan consisting of definitive or palliative radiation therapy and/or chemotherapy with or without surgery.

* Negative urine pregnancy test if a woman of child-bearing potential (WOCBP).
* WOCBP must be using an adequate method of contraception to avoid pregnancy throughout the study period.
* All patients will be evaluated in a uniform manner at the Stanford GI Combined Modality Tumor Board to determine eligibility. Exclusion Criteria:1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

  2. Any concurrent malignancy other than non-melanomaskin cancer, or carcinomainsitu of the cervix. Patients with a previous malignancy without evidence of disease for >5 years will be allowed to enter the trial.

  3. WOCBP who is pregnant or breastfeeding. 4. Inability to sign written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the performance of the novel imaging methods

SECONDARY OUTCOMES:
Correlate FLT activity with clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Albert Koong, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States